CLINICAL TRIAL: NCT01071343
Title: Effect of Transcutaneous Electric Muscle Stimulation on Muscle Volume in Patients With Septic Shock
Brief Title: Transcutaneous Electric Muscle Stimulation (TEMS) in Septic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Jesper Brøndum Poulsen, MD, Rigshospitalet, University of Copenhagen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H-KF-283379
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-01

CONDITIONS: Septic Shock
Keywords: muscular atrophy; recovery of function; rehabilitation; Intensive care unit
MeSH Terms: conditions — Shock, Septic; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transcutaneous electrical muscle stimulation — After randomization of the quadriceps muscles TEMS is applied on the intervention side for 7 consecutive days, 60 minutes per day.

SUMMARY:
A growing number of critically ill patients survive intensive care to be discharged from hospital. However, critical illness and prolonged bedrest are associated with muscle wasting with subsequent implications for recovery of normal physical function. Thus, one year after discharge, survivors of septic shock have reported prolonged and severe impairment of physical function.

Early interventions employed in the ICU to counteract loss of muscle mass may potentially improve physical outcome and reduce the overall burden of critical illness. As a potential supplement to physical therapy, transcutaneous electric muscle stimulation (TEMS) is a non-invasive method directed at maintaining skeletal muscle function through artificially induced contractions that are independent of patient efforts. TEMS has previously proven effective at preventing loss of muscle mass and force in a number of non-ICU patient groups, but has only been assessed sparsely in an ICU population where both immobilisation and systemic inflammation are present.

Therefore, the aim of the present study was to assess the effect of early TEMS on muscle volume in patients admitted to the intensive care unit with septic shock. The investigators hypothesized that this intervention would preserve muscle volume during septic shock.

DETAILED DESCRIPTION:
To ensures baseline comparability, eliminates many of the inter-individual confounding factors often present in ICU patients and enhances statistical strength we designed a study where we included a well-defined group of patients with septic shock in a single-legged exercise design, using the contralateral leg as the (paired) control and used a two-channel stimulation approach with 3-D evaluation of muscle volume changes based on CT scans.

After randomization of the quadriceps muscles TEMS is applied on the intervention side for 7 consecutive days, 60 minutes per day. All patients undergoes CT scans of both thighs before and immediately after the 7-day treatment period. The quadriceps muscle is then manually delineated on the transverse CT slices, and muscle volumes are calculated after 3-D reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients with septic shock admitted to the ICU of Rigshospitalet
* written informed consent from patient or proxy

Exclusion Criteria:

* diabetes
* a focus of infection in or trauma to the lower extremities
* a predicted ICU stay of less than seven days
* severe respiratory or circulatory instability that precluded transportation of the patient to the CT scanner
* patients receiving hihg dose corticosteroids (equivalent to methylprednisolone 1mg/kg/day or more)
* pregnancy
* severe psychiatric disorder
* > 72 hours since the diagnosis of septic shock was established
* > 7 days immobilisation prior to time of inclusion
* patient receiving neuromuscular blocking agents
* pre-existing neuromuscular disease
* acute compression/affection of central or peripheral nerves relevant to the lower extremities
* BMI > 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Volume of quadriceps muscles were calculated after 3-D reconstruction based on CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Jesper B Poulsen, MD, Principal Investigator — Rigshospitalet, University of Copenhagen; Kirsten Møller, MD, PhD, DMSci, Study Chair — Rigshospitalet, University of Copenhagen; Anders Perner, MD, PhD, Study Chair — Rigshospitalet, University of Copenhagen; Henrik Kehlet, MD, DMSci, Study Chair — Rigshospitalet, University of Copenhagen
Locations (1):
- Dept. of Intensive Care, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark